CLINICAL TRIAL: NCT01504425
Title: An Observational Study of Difficult Colonic Polypectomies
Brief Title: Difficult Colon Polypectomies
Status: Completed | Type: Observational
Sponsor: Clinical Hospital Colentina (Other)
Responsible Party: Principal Investigator, dr. Theodor Alexandru Voiosu, MD, Clinical Hospital Colentina
Other Study IDs: COL-GASTRO-1
Record Dates: First submitted 2012-01-03; First posted 2012-01-05 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Colon Polyps
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The investigators aim to define the concept of difficult colonic polypectomy and investigate whether resection methods (hot/cold snare, Endoscopic mucosal resection (EMR), endoscopic submucosal dissection (ESD)), adjuvant techniques (endoloop, prophylactic hemoclip placement, submucosal injection) and operator experience have an impact on polypectomy outcomes and complication rate.

ELIGIBILITY:
Inclusion Criteria:

* colonic polyps that are deemed difficult to resect by the endoscopist

Exclusion Criteria:

* patient refusal to participate in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with colonic polyps that are deemed difficult to resect
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2011-12; Primary Completion 2013-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
complication rate | 30 days
  the advent of hemorrhage or perforation during the 30 days following the endoscopic procedure

CONTACTS AND LOCATIONS:
Overall Officials: Theodor Voiosu, MD, Principal Investigator — Clinical Hospital Colentina
Locations (1):
- Colentina Hospital, Bucharest, Romania

REFERENCES:
- [Result] Voiosu T, Ratiu I, Hervoso CM, Furnari M, Voiosu A, Goldis A, Mateescu B, Tacconi M, Dulbecco P, Haidar A, Voiosu MR, Sporea I. Polyp and endoscopist-related factors influencing complication rates in difficult colonic polypectomies: results of a multicenter observational study. Rom J Intern Med. 2013 Jul-Dec;51(3-4):172-8. PMID 24620630